CLINICAL TRIAL: NCT04162639
Title: The Relationship Between Cadaveric Allograft Skin and Human-leukocyte Antigens (HLA)-Sensitivity in Burn Patients
Brief Title: The Relationship Between Cadaveric Allograft Skin and HLA-Sensitivity in Burn Patients
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: PI is working on getting funding for the study and wishes to withdraw the study until that funding is secured.
Sponsor: Virginia Commonwealth University (Other)
Collaborators: AlloSource (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: HM20015249
Record Dates: First submitted 2019-11-11; First posted 2019-11-14 (Actual); Last update posted 2021-03-19 (Actual); Status verified 2021-03

CONDITIONS: Burns
MeSH Terms: conditions — Burns

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- One donor (Experimental): Participants will receive skin allograft from 1 distinct cadavers.
  Interventions: Biological: Skin allograft
- Two donors (Experimental): Participants will receive skin allograft from 2 distinct cadavers.
  Interventions: Biological: Skin allograft
- Three donors (Experimental): Participants will receive skin allograft from 3 distinct cadavers.
  Interventions: Biological: Skin allograft
- Control (No Intervention): Participants will be burned patients with wounds that do not require skin allografts, but are instead reconstructed with their own skin (skin autografts) in a single stage.

INTERVENTIONS:
Biological: Skin allograft — Participants will receive skin allograft from either 1, 2 or 3 distinct cadavers. This skin allograft will be applied in a routine fashion, with no deviation from the typical clinical course of treatment.
  Arms: One donor; Three donors; Two donors

SUMMARY:
The purpose of this research study is to look at how the body's immune system reacts to temporary skin grafts from deceased donors.

DETAILED DESCRIPTION:
Some burns will heal best with the use of temporary skin grafts from cadavers before covering the burns with grafts of the patient's own skin. This is the usual care for these types of burn injuries recommended by burn surgeons. This skin is applied in the operating room and removed after several days. During that time, the body's immune system will make antibodies to the skin. Normally, these antibodies are harmless. However, extra antibodies can make it difficult to find donors for transplants. The results of this study will be used to better understand how to treat a subset of burn patients with very severe burns in a way that allows them to receive tissue transplants (e.g. face transplants, hand transplants).

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years or older
* Burns of deep partial thickness or full thickness depth totaling less than or equal to 10% total body surface area.
* Injury requiring staged reconstruction with allograft skin (experimental group)
* Injury requiring reconstruction with autograft skin (i.e. no cadaver skin; control group)

Exclusion Criteria:

* Burns exceeding 10% total body surface area.
* Pre-existing allosensitization at time of injury
* Blood or blood product transfusion requirement
* Pregnancy at the time of injury or during study period
* History of solid organ transplant during study period
* History of autoimmune disorder (systemic lupus erythematosus, etc.)
* History of mechanical circulatory support (extracorporeal membrane oxygenation, ventricular assist device, total artificial heart) during study period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-02 (Estimated); Primary Completion 2023-02 (Estimated); Study Completion 2023-02 (Estimated)

PRIMARY OUTCOMES:
Change in participant's panel reactive antibody (PRA) score at 1 month | Baseline to 1 month
  Standard PRA assays will be performed on blood samples drawn from participants giving a percent score representing the number of reactions in the sample.
Change in participant's panel reactive antibody (PRA) score at 6 months | Baseline to 6 months
  Standard PRA assays will be performed on blood samples drawn from participants giving a percent score representing the number of reactions in the sample.
Change in participant's panel reactive antibody (PRA) score at 12 month | Baseline to 12 months
  Standard PRA assays will be performed on blood samples drawn from participants giving a percent score representing the number of reactions in the sample.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Feldman, Principal Investigator — Virginia Commonwealth University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Duhamel P, Suberbielle C, Grimbert P, Leclerc T, Jacquelinet C, Audry B, Bargues L, Charron D, Bey E, Lantieri L, Hivelin M. Anti-HLA sensitization in extensively burned patients: extent, associated factors, and reduction in potential access to vascularized composite allotransplantation. Transpl Int. 2015 May;28(5):582-93. doi: 10.1111/tri.12540. Epub 2015 Feb 26. PMID 25683513
- [Background] Klein HJ, Lehner F, Schweizer R, Rusi-Elsener B, Nilsson J, Plock JA. Screening of HLA sensitization during acute burn care. Burns. 2018 Aug;44(5):1330-1335. doi: 10.1016/j.burns.2018.01.010. Epub 2018 Mar 7. PMID 29929900
- [Background] Klein HJ, Schanz U, Hivelin M, Waldner M, Koljonen V, Guggenheim M, Giovanoli P, Gorantla VS, Fehr T, Plock JA. Sensitization and desensitization of burn patients as potential candidates for vascularized composite allotransplantation. Burns. 2016 Mar;42(2):246-57. doi: 10.1016/j.burns.2015.05.019. Epub 2015 Sep 29. PMID 26392022